CLINICAL TRIAL: NCT05321030
Title: Correlation Between Smartphone Addiction and Back Dysfunction and Core Muscle Morphology and Performance in Asymptomatic Young Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Hussin, Principal investigator, Cairo University
Other Study IDs: Asmaa_PhD_2022
Record Dates: First submitted 2022-03-19; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Back Disorder; Smartphone Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smartphone addict
- Smartphone non addict

SUMMARY:
The purpose of this study is to investigate the association between smartphone addiction and back pain, function, and lumbar stabilizer cross-sectional area and thickness compared with non-addicted teenagers.

DETAILED DESCRIPTION:
Smartphone prolonged use has been suggested as a risk factor for psychological, visual, and musculoskeletal dysfunctions. The musculoskeletal dysfunction may be related to direct contact use with smartphones as in thumb, elbow, and neck pain. Moreover, indirect long use of smartphones may affect thoracic, lumbar, and lower limbs.

COVID-19 pandemic occurred in a time of outstanding scientific progress and global digitalization. Therefore, smartphone usage became a must for human connection, learning, and entertainment, providing psychological and social support. In the meantime, it was observed a significant increase in overuse and addiction, especially in young and teenage females. The addiction is associated with more musculoskeletal abnormalities when compared to non-addict users. Several studies found an association between smartphone usage and back pain, concomitant with a reduction in thoracic extensors activity. This back pain may affect their quality of life and work-related productivity. However, the relationship between back dysfunction and smartphone addiction is still unclear. A few attempts were done to elucidate this relationship. Yet if proven correct, then preventive measures such as recommendations and precautions regarding smartphone use could be distributed to users by the manufacturers. Furthermore, engineering solutions are needed to optimally design smartphones to alter their weight and sizes to minimize potential adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 years to 30 years.
2. BMI between 19.0-29.9 kg/m2.

Exclusion Criteria:

1- Previous history of spinal trauma or dysfunction. 2 - Any systemic disease that may affect spine such as ankylosing spondylitis and rheumatoid arthritis.

3 - Cognitive or memory impairment in memory or cognitive function.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Using G-power version 3.1.9.7 for windows and regarding T-test study, alpha level of 0.05, confidence interval 95% and effect size of 0.25 (to detect small effects), two groups and six dependent variables, the total sample size was 136 subjects.
Sampling Method: Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of back function and disability | at baseline only
  Functional disability will be assessed by the Oswestry disability questionnaire, a functional scale assessing the impact of LBP on daily activities. It is a self-administered, 10-item questionnaire: the first section rates the intensity of pain and the others describe its disabling effect on typical daily activities. The score for each item ranges from 0 to 5, the score is calculated by the addition of the values assigned for each of the 10 individual questions
Musculoskeletal assessment By Ultrasonography | at baseline only
  Ultrasonography will be used for measuring CSA and MT of LMM. Muscle thickness measurement by US.
Core muscles strength | at baseline only
  Core stability will be measured using prone and supine bridging as bridging maneuvers seem to be practical, reliable, and valid methods of reflecting lumbar spine stabilization endurance capability. In prone bridge each subject will be in the prone position, supporting on the elbows. The elbows will be spaced shoulder-width apart, and the feet were set with a narrow base, but not touching. The subject then asked to raise the pelvis from the floor so that only the forearms and the toes were in contact with the floor. The shoulders, hips, and ankles were maintained in a straight line.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Hussin, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided